CLINICAL TRIAL: NCT05976516
Title: Study on the Correlation Between CXCL2/CXCL8 and the Degree of Intervertebral Disc Degeneration and Radiological Progress
Brief Title: CXCL2/CXCL8 Promote Intervertebral Disc Degeneration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, pengfei, xue, Dr, Zhongda Hospital
Other Study IDs: 20220224016
Record Dates: First submitted 2023-02-19; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Cytokine; Intervertebral Disc, Degenerative
Keywords: cytokine; chemokine; Intervertebral Disc Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- pirffmann 2 grade
  Interventions: Diagnostic Test: CXCL2/CXCL8
- pirffmann 3 grade
  Interventions: Diagnostic Test: CXCL2/CXCL8
- pirffmann 4 grade
  Interventions: Diagnostic Test: CXCL2/CXCL8
- pirffmann 5 grade
  Interventions: Diagnostic Test: CXCL2/CXCL8

INTERVENTIONS:
Diagnostic Test: CXCL2/CXCL8 — Detecte CXCL2/8 content in nucleus pulposus and peripheral blood of patients in each group

SUMMARY:
Low back pain (LBP) is the largest cause of morbidity in the world, and about 80% of Chinese people are affected in their lifetime. Although the prevalence of IDD gradually increases with age, IDD is very common among subjects under 30 years old. In addition to age, there are other factors, such as excessive or uneven mechanical load, obesity, genetics, nutrition, trauma and gender. In addition, it is not clear whether the heavy physical load associated with occupation is an important risk factor for IDD. Some studies have found that IDD is more common among athletes than the general population. Due to the complexity and multifactorial nature of IDD, its pathogenesis and risk factors are still unclear, which seriously hinders the rational stratification of LBP patients and limits the development of personalized treatment.

ELIGIBILITY:
Inclusion Criteria:

* It meets the diagnostic criteria of lumbar disc degeneration; No previous history of spinal surgery; Good ability of independent behavior and cooperation in completing research; The patient is aware of this study and has signed the consent form.

Exclusion Criteria:

* Patients with spinal tumor, infection, tuberculosis and other diseases; Patients with claustrophobia; Parkinson's syndrome patients; Poor cooperation, Poor image quality; Patients with osteoporosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with lumbar disc herniation who went to the spinal surgery department of Zhongda Hospital
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
CXCL2/8 content | 1 month
  CXCL2/CXCL8 content of nucleus pulposus

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No